CLINICAL TRIAL: NCT05805540
Title: Acute Effects on Creatine Kinase, Perceived Fatigue and Physical Performance of Different Post-Exercise Recovery Methods in Elite Basketball Players: A Crossover Randomized Controlled Trial
Brief Title: Effects on CK, RPE, VAS Scale and Physical Performance of Three Recovery Methods in Elite Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: The RECOVERY Study
Record Dates: First submitted 2023-03-27; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Cold-water Immersion; Protein-carbohydrates Supplementation; Active Recovery; Placebo
Keywords: cryotherapy; recovery strategies; nutrition; team sports; invisible training; exercise-induced muscle damage

STUDY DESIGN:
Intervention Model Description: A crossover design was used to examine the effects of four different recovery interventions on muscle damage and fatigue and physical performance after a maximal exercise test in elite male basketball players. Thus each athlete performed all the recovery methods that were included in the study, one week apart; including CWI, carbohydrate-protein supplementation, active recovery, and placebo-control condition.
Who Masked: Participant, Investigator
Masking Description: Both the participants and the investigators who performed the intervention were didn't know whether they were drinking the protein-carbohydrate supplementation or the placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold-water immersion (Experimental): Subjects were immersed, in a sitting position where legs were always covered, in cold water at 11ºC in periods of 2 minutes submerged and 2 minutes out of the water at room temperature (25ºC), repeating this process 5 times.
  Interventions: Procedure: Cold-water immersion
- Protein-carbohydrates supplementation (Experimental): Subjects consumed a mixed carbohydrate and protein beverage, composed of 0.3gr/kg of maltodextrin and 0.2gr/kg of neutral whey protein in 0.5 litres of water.
  Interventions: Procedure: Protein-carbohydrates supplementation
- Active recovery (Experimental): Subjects was carried out using a bicycle ergometer. The subjects pedaled for 25 minutes at 50% of the maximum heart rate (HRmax).
  Interventions: Procedure: Active recovery
- Placebo (Placebo Comparator): Subjects drank a water-based drink and sweetener. Both the PLA and SUPPL group sat for 25 minutes until all recovery methods were completed.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Cold-water immersion — Subjects were immersed, in a sitting position where legs were always covered, in cold water at 11ºC in periods of 2 minutes submerged and 2 minutes out of the water at room temperature (25ºC), repeating this process 5 times
  Arms: Cold-water immersion
Procedure: Protein-carbohydrates supplementation — Subjects consumed a mixed carbohydrate and protein beverage, composed of 0.3gr/kg of maltodextrin and 0.2gr/kg of neutral whey protein in 0.5 litres of water. Subject sat for 25 minutes until all recovery methods were completed.
  Arms: Protein-carbohydrates supplementation
Procedure: Active recovery — Subjects was carried out using a bicycle ergometer. The subjects pedaled for 25 minutes at 50% of the maximum heart rate (HRmax)
  Arms: Active recovery
Procedure: Placebo — Subjects drank a water-based drink and sweetener. Subject sat for 25 minutes until all recovery methods were completed.
  Arms: Placebo

SUMMARY:
The aim of this study was to compare the effects of cold water intermittent ion (CWI), carbohydrate and protein supplementation (SUPPL), and active recovery (ACT) on creatine kinase (CK), perceptual and performance markers of recovery in elite basketball players after a specific fatigue protocol.

Fifteen elite basketball players participated in this crossover controlled trial. All participants were randomly measured in 4 conditions of the recovery method 1 week apart after a fatigue exercise protocol (~ 45 'of high intensity intermittent effort with specific basketball movements). The recovery methods consist of CWI at 10oC in periods of 2 minutes submerged and 2 minutes out of the water, supplementation with 0.3gr / kg of maltodextrin and 0.2gr / kg of neutral whey protein in 0.5 liters of water, pedaling ACT for 25 minutes at 50% of maximum heart rate or a placebo drink (PLA). The Visual Analogue Fatigue Scale (VAS), Perceived Exercise Rate (RPE), CK and physical performance (jumping, speed, isometric and dynamic tests of resistance to squats) were measured before, after and 24 hours after of the protocol. The VAS scale and RPE were also measured immediately after application of the recovery method. Repeated 2-way post-hoc comparisons of ANOVA and Bonferroni measures were applied, with a significance set at P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Having at least 10 years of sports practice,
* Having been training during the season a minimum of four times a week,
* Not having suffered serious or minor but recently injuries,
* Having competed and trained regularly in the previous season.

Exclusion Criteria:

* Suffering an injury during the study period
* Not having gone through all the treatment groups (CWI, carbohydrate-protein supplementation, active recovery and placebo)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Creatine Kinase (CK) | 4 Weeks
  Blood samples were obtained from the earlobe and collected into capillary tubes. Serum creatine kinase activity was analyzed with Reflotron ® Plus - Roche
Fatigue perception | 4 Weeks
  The VAS fatigue scale (VAS) was used and evaluated on a scale from 1 to 10 (1 = no fatigue and 10 = extremely fatigued).
Rate of Perceived Exertion | 4 Weeks
  The Rate of Perceived Exertion Scale (RPE) was used and evaluated on a scale from 1 to 10 (1 = no exertion and 10 = extremely hard).
10 meters sprint time | 4 Weeks
  10m Sprint Test was used and subjects ran 10m maximally. The subjects had 2 attempts to achieve their best performance with 1 minute of rest between trials. Time was recorded with a video analysis.
4 x 10 meters agility time | 4 Weeks
  4 x 10m Agility Test was used and subjects had to run as fast as possible between two cones 10 meters apart four times. The subjects had 2 attempts to achieve their best performance with 1 minute of rest between trials. Time was recorded with a video analysis.
Squat Jump | 4 Weeks
  The flight time in jumps height and its maximal speed were used as a measure of maximal muscle power and was measured on a force platform (Quattro Jump, Kristler). In squat jump, the subjects were asked to keep their hands on their hips and beginning the jump with a 90º knee flexion, without countermovement. Subjects had 2 attempts to achieve their best jump with 3 minutes of rest between trials.
Counter Movement Jump | 4 Weeks
  The flight time in jumps height and its maximal speed were used as a measure of maximal muscle power and was measured on a force platform (Quattro Jump, Kristler). In countermovement jump, subjects were only asked to keep their hands on their hips and jump as high as possible, with countermovement. Subjects had 2 attempts to achieve their best jump with 3 minutes of rest between trials.
Abalakov Jump | 4 Weeks
  The flight time in jumps height and its maximal speed were used as a measure of maximal muscle power and was measured on a force platform (Quattro Jump, Kristler). Abalakov jump was performed with free arms movement and countermovement. Subjects had 2 attempts to achieve their best jump with 3 minutes of rest between trials.
Half Squat Isometric Strength | 4 Weeks
  In the maximal isometric strength test, the subjects performed a maximal isometric contraction in the half squat exercise, with 90º knee flexion. The strength of the subjects was measured with a force platform on which the exercise was performed. The subjects were asked to perform the maximal strength possible since the start and to not stop until a signal. They had 2 attempts to achieve their best performance with 3 minutes of rest between trials.
Half Squat Dynamic Strength | 4 Weeks
  In the dynamic strength test, the subjects performed 6 repetitions of a half squat, using a Smith Machine, with the load that represented the 70% of RM (0.65 m·s) at baseline in the half squat exercise. The mean velocity was measured with a linear encoder and it was registered the fastest repetition. The subjects were asked to perform the concentric action as fast as possible. They had 2 attempts to achieve their best performance with 3 minutes of rest between trials.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús G Ponce, PhD, Principal Investigator — University of Cádiz
Locations (1):
- Science of Education Faculty, Puerto Real, Cadiz, Spain